CLINICAL TRIAL: NCT02147288
Title: Prevention of Seroma Formation and Wound Complications Using NPWT Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIC# 1010007535
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Seroma; Wound Dehiscence; Wound Infection
MeSH Terms: conditions — Seroma; Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Breast Recon with acellular dermal matrix (ADM) on NPWT (Experimental)
  Interventions: Device: Renasys*GO Negative Pressure Wound Therapy System
- Lipoabdominoplasty on NPWT (Experimental): The Smith&Nephew Renasys*GO device connected to non-compressible drains will be applied to the lipoabdominoplasty patients enrolled in this arm.
  Interventions: Device: Renasys*GO Negative Pressure Wound Therapy System
- Abdominoplasty on NPWT (Experimental): The Smith&Nephew Renasys*GO device connected to non-compressible drains will be applied to the abdominoplasty patients enrolled in this arm.
  Interventions: Device: Renasys*GO Negative Pressure Wound Therapy System
- Ventral Hernia Repair (VHR) on NPWT (Experimental): The Smith&Nephew Renasys*GO device connected to non-compressible drains will be applied to the VHR patients enrolled in this arm.
  Interventions: Device: Renasys*GO Negative Pressure Wound Therapy System
- Panniculectomy on NPWT (Experimental): The Smith&Nephew Renasys*GO device connected to non-compressible drains will be applied to the panniculectomy patients enrolled in this arm.
  Interventions: Device: Renasys*GO Negative Pressure Wound Therapy System
- Breast Recon with ADM on Jackson-Pratt (JP) Drains (No Intervention): Standard of Care. The Jackson-Pratt (JP) drain is used following surgery to collect bodily fluids from the surgical site.
- Abdominoplasty on JP Drains (No Intervention): Standard of Care. The Jackson-Pratt (JP) drain is used following surgery to collect bodily fluids from the surgical site.
- Lipoabdominoplasty on JP Drains (No Intervention): Standard of Care. The Jackson-Pratt (JP) drain is used following surgery to collect bodily fluids from the surgical site.
- Ventral Hernia Repair (VHR) on JP Drains (No Intervention): Standard of Care
- Panniculectomy on JP Drains (No Intervention): Standard of care. The Jackson-Pratt (JP) drain is used following surgery to collect bodily fluids from the surgical site.

INTERVENTIONS:
Device: Renasys*GO Negative Pressure Wound Therapy System — Continuous, mechanical negative pressure wound therapy applied to drain in the immediate post-operative period (vs standard, closed-suction JP drains).
  Other Names: Smith & Nephew, Inc.
  Arms: Abdominoplasty on NPWT; Breast Recon with acellular dermal matrix (ADM) on NPWT; Lipoabdominoplasty on NPWT; Panniculectomy on NPWT; Ventral Hernia Repair (VHR) on NPWT

SUMMARY:
The specific aim of this study is to improve post-operative wound care in the morbidly-obese body-contouring patient population following massive weight loss undergoing either panniculectomy or formal abdominoplasty, those patients undergoing complex abdominal wall reconstruction (i.e. ventral hernia repair) and breast reconstruction with acellular dermal matrix, as well as patients undergoing regular lipo-abdominoplasty by comparing the effectiveness of standard closed-suction drains versus the immediate application of continuous negative pressure via a NPWT (negative pressure wound therapy) device attached to non-compressible drains. Additionally, we aim to demonstrate increases both in cost-effectiveness and quality of life in these patients with the use of the NPWT wound care apparatus.

Hypothesis 1 Continuous negative pressure devices decrease the incidence of wound complications in comparison with conventional closed suction drains when used in patients after massive weight loss undergoing body-contouring procedures (panniculectomies alone and formal abdominoplasties), and in patients undergoing VHR and breast reconstruction with acellular dermal matrix, as well as those undergoing regular lipo-abdominoplasty.

Hypothesis 2 Although initially more costly than traditional closed suction drains, the use of continuous negative pressure devices will in the long-term result in lower total health care costs in the above-stated patient population due to a decreased need for additional procedures and/or clinical management, including surgical interventions, hospital admissions, administration of antibiotics, multiple follow-up office visits, and chronic wound care.

Hypothesis 3 Better quality of life is associated with the use of continuous negative pressure devices compared to closed suction drains in these patient populations.

DETAILED DESCRIPTION:
In collaboration with the Yale Bariatric Surgery Program and General Surgery Department, patients will be identified as 18-years-of-age or older seeking body-contouring procedures (including panniculectomy and abdominoplasty) following massive weight loss or those patients in need of complex abdominal wall reconstruction (i.e. ventral hernia repair) and breast reconstruction necessitating the use of acellular dermal matrix. For the timeframe outlined in this protocol, the Section of Plastic Surgery at Yale performs surgeries in excess of the required numbers needed for this study, ensuring timely completion.

Exclusion criteria will include the FDA-identified contraindications to use of continuous negative pressure suction devices, as follows:

* presence of necrotic tissue
* untreated osteomyelitis
* malignancy (except terminal patients for quality of life issues)
* untreated malnutrition
* use on exposed arteries, veins, or organs
* use on non-enteric and unexplored fistulas Special precaution will be taken when using the NPWT device in patients on anticoagulants, exhibiting otherwise difficult hemostasis, or non-adherent patients.

Following a detailed explanation of the study design as well as the associated risks and benefits that may be incurred by each potential test group, patients who agree to participate in the study (via informed consent) will be categorized by characteristics including past medical history, past surgical history, social history, pre- and post-bariatric surgery total weight loss and BMI and will be randomized into either the control (standard closed suction drains) or experimental (continuous negative pressure via NPWT device) arm of each group, depending on the procedure to be performed, as follows:

1. 30 total patients undergoing panniculectomy alone following massive weight loss
2. 30 total patients undergoing formal abdominoplasty (including undermining of skin flaps, rectus fascia plication and liposuction) following massive weight loss
3. 30 total non-massive weight loss patients undergoing formal lipo-abdominoplasty
4. 30 total patients undergoing ventral hernia repair using acellular dermal matrix
5. 30 total patients undergoing bilateral breast reconstruction using acellular dermal matrix with 30 breasts randomized to conventional closed suction (one breast left vs right) and 30 breasts randomized to continuous negative pressure devices (=60 breasts total)

The control subject arm of each procedure group will be outfitted with 2 standard closed suction Jackson-Pratt (JP) drains for a period of 4 weeks (unless otherwise specified by the principle investigator at the point of follow-up), both as an inpatient and at home. The experimental subject arm of each procedure group will be outfitted with 2 non-compressible Blake drains attached to continuous suction via NPWT device for a period of 4 weeks (unless otherwise specified by the principle investigator at the point of follow-up), both as an inpatient and at home.

In the breast reconstruction group there will be an internal control via the 30 breasts drained conventionally in the same patient.

To achieve better control of variables, the total length of the incision and area of skin- undermining along the midline will also be measured and documented in the massive weight loss patient group to:

1. exactly distinguish the formal abdominoplasty from the panniculectomy patients and
2. evaluate to what extent skin-undermining is a contributing factor to seroma-formation compared to the patients' intrinsic factors.

All patients from group 1 will be wearing compression girdles starting post-operative day #1; patients from groups 2 and 3 will start wearing the compression girdles post-operative day #7 (to minimize the risk of central skin flap necrosis); and patients in group 4 will start wearing a regular abdominal binder on post-operative day #1.

The amount of tumescent solution as well as the amount of lipo-aspirate will be recorded in each patient in groups 2 & 3.

The following chart will be provided for follow-up lab studies and clinic visits:

Wound-Healing Research Study Schedule and Logistics

Post-Op Follow-up Activities *Duration Week 1 Formal Outpatient Clinic Visit 30 minutes Follow-Up Blood Labs #1 15 minutes Quality of Life Survey #1 30 minutes

Week 2 Formal Outpatient Clinic Visit 30 minutes Follow-up Blood Labs #2 15 minutes Ultrasound Examination #1 15-30 minutes

Week 3 Ultrasound Examination #2 15-30 minutes (No formal clinic visit)

Week 4 Formal Outpatient Clinic Visit 30 minutes Quality of Life Survey #4 30 minutes

Week 8 Formal Outpatient Clinic Visit 30 minutes

*All visit duration times are approximate.

Per routine post-operative protocols, patients will be seen in clinic at week 1, 2, 4, and 8, and as needed clinically. Ultrasounds will be performed for research purposes only at the 2nd and 4th week visits, and diagnostically in the event that complications arise at any other point during the post-operative period. QALY surveys will be performed at the 1st and 4th week post-operative clinic visits.

Together with standard pre-operative blood work, (i.e., complete blood count (CBC), basic electrolyte panel, International Normalized Ratio (INR)/prothrombin time test (PT)/partial thromboplastin test (PTT)), we will also obtain albumin, pre-albumin and total protein levels in each patient on post operative days (PODs) #7 and #14.

Outcomes will be measured as follows:

* Total amount of fluid drainage comparing the two systems at 1, 2, 4, and 8 weeks (as long as drains remain in place)
* Analysis of complication rates including the incidence of infection requiring antibiotics, wound dehiscence, and the need for seroma drainage and/or surgical revision.
* Quantification of seroma formation by ultrasound examination of 5 regions of the abdominal wall: epigastrium (EPI), umbilical (UMB), hypogastrium (HYPO), right iliac fossa (RIF) and left iliac fossa (LIF)], at two postoperative periods: (P1), between postoperative days #11 and #14, and (P2), between postoperative days #18 and #21 as described by DiMartino et al [20], as well as ultrasound of the superior, medial, lateral and inferior portions of the reconstructed breasts.

Subjects included in the control (standard closed suction drains) and experimental arms (NPWT device) of each procedure group will not experience risks to subject privacy, discomforts, or inconveniences associated with participating in this research project that they would not otherwise experience with the use of standard closed suction drains currently being used for post-operative wound care. These standard risks, discomforts, and inconveniences include the potential for bleeding from drain site, infection at drain site, requirement of changing collection vessel when full, and pain. The post-operative ultrasound evaluation is also non-invasive. It is an evaluation which is often performed on patients in the post-operative period to assess for subcutaneous fluid collections.

The cost-effectiveness of each approach to post-surgical drain placement and design will be assessed via tracking patient health care costs associated with the specific surgical procedure performed, the costs associated with immediate post-surgical care, and any follow-up care incurred during the prolonged post-operative period as designated in the study design. The relevant costs will be compared between the control and experimental groups of each arm of the study and the cost-effectiveness ratio will be calculated using an objective, validated quality of life assessment.

Quality of life will be assessed via an incremental cost-effectiveness ratio, namely the repeatedly validated quality adjusted life year (QALY) metric achieved through patient surveys/interviews. The dynamic health assessment survey (DYNHA SF-36) will be used to evaluate patient health outcomes.

The DYNHA SF-36 Health Survey is a computerized adaptive testing (CAT) version of the industry standard, fixed-length Short Form Health Survey (SF-36) that has been translated and made available for use in many country and language-based cohorts [21]. The SF-36 focuses on assessing functional health and well-being, measuring eight health domains, including physical functioning, bodily pain, the ability to engage in work and leisure activities, psychological distress, vitality, and emotional health in order to accurately evaluate an individual's physical and mental status throughout the recovery period. The advantages of a dynamic health assessment include brevity without sacrificing accuracy, a focus on parameters affected by chronic health conditions, reliable outcomes for monitoring individuals, lower data collection costs, and real-time results with built-in interpretation and scoring.

Regarding the breast reconstruction group, we do not feel that by employing two different techniques (i.e. continuous vs intermittent/ bulb suction) in the same patient this would lead to a psychological burden for the patient. We expect that the main outcome difference in this group will be regarding the ease and comfort with the continuous suction device over the standard bulb suction. While the patients will likely prefer one over the other device, this should not have tremendous impact on their recovery in general or in how they cope with their disease.

ELIGIBILITY:
Inclusion Criteria:

* 30 total patients undergoing panniculectomy alone following massive weight loss
* 30 total patients undergoing formal abdominoplasty (including undermining of skin flaps, rectus fascia plication and liposuction) following massive weight loss
* 30 total non-massive weight loss patients undergoing formal lipo-abdominoplasty
* 30 total patients undergoing ventral hernia repair using acellular dermal matrix
* 30 total patients undergoing bilateral breast reconstruction using acellular dermal matrix with 30 breasts randomized to conventional closed suction (one breast left vs right) and 30 breasts randomized to continuous negative pressure devices (=60 breasts total)

Exclusion Criteria:

* presence of necrotic tissue
* untreated osteomyelitis
* malignancy (except terminal patients for quality of life issues)
* untreated malnutrition
* use on exposed arteries, veins, or organs
* use on non-enteric and unexplored fistulas Special precaution will be taken when using the NPWT device in patients on anticoagulants, exhibiting otherwise difficult hemostasis, or non-adherent patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J G Thomson, MD, Principal Investigator — Section of Plastic and Reconstructive Surgery, Department of Surgery, Yale University School of Medicine
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Walker ME, Tsay C, Broer PN, Zhu VZ, Sturrock T, Ng R, Scoutt LM, Thomson JG, Kwei SL. A prospective, randomized-controlled pilot study comparing closed suction versus negative pressure drains for panniculectomy patients. J Plast Reconstr Aesthet Surg. 2018 Mar;71(3):438-439. doi: 10.1016/j.bjps.2017.11.013. Epub 2017 Nov 28. No abstract available. PMID 29289501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited for the "panniculectomy on negative pressure wound therapy (NPWT)" and "panniculectomy on Jackson-Pratt (JP) drains" groups. Patients were not recruited for the remaining arm;s the manufacturer, Smith & Nephew, temporarily halted on the distribution of the device (Renasys*GO negative pressure wound management system).
Groups:
- Panniculectomy on Jackson Pratt (JP) Drains: Standard of Care
- Panniculectomy on Negative Pressure Wound Therapy (NPWT): The Smith&Nephew Renasys*GO device connected to non-compressible drains will be applied to the panniculectomy patients enrolled in this arm.
  Renasys*GO Negative Pressure Wound Therapy System: Continuous, mechanical negative pressure wound therapy applied to drain in the immediate post-operative period (vs standard, closed-suction JP drains).
Period: Overall Study
Arm/Group | Panniculectomy on Jackson Pratt (JP) Drains | Panniculectomy on Negative Pressure Wound Therapy (NPWT) | Breast Recon With Acellular Dermal Matrix (ADM) on NPWT | Breast Recon With ADM on Jackson-Pratt (JP) Drains | Lipoabdominoplasty on NPWT | Lipoabdominoplasty on JP Drains | Abdominoplasty on NPWT | Abdominoplasty on JP Drains | Ventral Hernia Repair (VHR) on NPWT | Ventral Hernia Repair (VHR) on JP Drains
Started | 22 | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 21 | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — post-operative hematoma | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — complications from concurrent hernia rep | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panniculectomy on JP Drains: Standard of Care
- Total: Total of all reporting groups
Arm/Group | Panniculectomy on JP Drains | Panniculectomy on NPWT | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Full Range); unit: years] | 41 [24 to 58] | 46 [26 to 65] | 43.6 [24 to 65]
Gender [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 3 | 1 | 4
Diabetes history [Number; unit: participants]
  diabetic | 6 | 3 | 9
  non-diabetic | 15 | 19 | 34
Smoking status [Number; unit: participants]
  smokers | 3 | 4 | 7
  non-smokers | 18 | 18 | 36
Prior abdominal surgery [Number; unit: participants]
  yes | 15 | 19 | 34
  no | 6 | 3 | 9
Body mass Index [Mean (Full Range); unit: kg/m^2] | 32.3 [23.1 to 49.1] | 30.4 [25.1 to 42.0] | 31.32 [23.1 to 49.1]
Pre-operative prealbumin [Mean (Full Range); unit: milligrams per deciliter] | 20.3 [8.9 to 34.6] | 21.4 [10.3 to 25.2] | 20.9 [8.9 to 34.6]
Incision length [Mean (Full Range); unit: centimeters] | 52.3 [26.0 to 96.0] | 56.6 [26.0 to 78.5] | 54.5 [26.0 to 96.0]
Specimen weight [Mean (Full Range); unit: kilograms] | 3.07 [0.74 to 8.52] | 2.61 [0.66 to 5.50] | 2.83 [0.66 to 8.52]
Drain duration [Mean (Full Range); unit: days] | 16 [8.0 to 25.0] | 14 [9.0 to 27.0] | 15 [8.0 to 27.0]

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Seroma Formation
Description: Quantitative assessment of fluid collection in pre-defined anatomic regions will be performed via ultrasound examination approximately two weeks following removal of drains (either JP or NPWT-associated)
Time Frame: Two weeks following drain removal
Population: Among 21 completers (standard of care group); one outlier was excluded from the analysis; 20 subjects were analyzed. Among 22 completers (experimental group), one outlier and 1 who did not have an ultrasound (i.e., fluid was not measured) were excluded, leaving 20 subjects for analysis.
Measure: Mean (Full Range); unit: cm^3
Arm/Group | Panniculectomy on JP Drains | Panniculectomy on NPWT
Number analyzed (Participants) | 20 | 20
cm^3 | 16.9 [0 to 132] | 10.1 [0 to 45.9]

ADVERSE EVENTS:
Arm/Group | Panniculectomy on JP Drains | Panniculectomy on NPWT
Serious Adverse Events (participants affected / at risk) | 1/22 | 2/24
Other Adverse Events (participants affected / at risk) | 7/22 | 4/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panniculectomy on JP Drains (N=22) | Panniculectomy on NPWT (N=24)
post-operative hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
abcess with infected mesh (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panniculectomy on JP Drains (N=22) | Panniculectomy on NPWT (N=24)
seroma (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
wound dehiscence (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
stitch absess (Skin and subcutaneous tissue disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes